CLINICAL TRIAL: NCT00117091
Title: An Open-Label Multicentre Study of Anakinra (Kineret®) in Combination With DMARDS in Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: Anakinra (Kineret®) in Combination With Disease Modifying Anti-Rheumatic Drugs (DMARDS) in Subjects With Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020364
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; Anakinra (Kineret®)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Drug: Anakinra (Kineret®)

SUMMARY:
The purpose of this study is to evaluate the percentage of subjects in Australian clinical practice continuing treatment with Anakinra (Kineret®) at the end of study week 48 in subjects with active RA. The continued use of Kineret® will be based on pre-defined response assessment criteria for subjects with active RA.

ELIGIBILITY:
Inclusion Criteria: - Subjects diagnosed with RA as determined by American College of Rheumatology (ACR) criteria with a disease duration of at least 24 weeks prior to enrollment - Active RA at screening as defined by EITHER: (1) At least 6 swollen joints (using a 66 joint count) and at least 6 tender joints (using a 68 joint count) OR (2) 4 non-hand joints and at least 1 of the following: *Morning stiffness of at least 45 minutes; *CRP greater than 1.5 mg/dL (15.0 mg/L); *ESR greater than 28 mm/h; *DAS28 greater than 3.2 - Subjects must have failed an adequate trial of at least 3 disease-modifying antirheumatic drugs (DMARDS) alone or in combination (one of which must be MTX) and have been on the same treatment and doses for 4 weeks prior to enrollment (i.e., an adequate trial is defined as 12 weeks unless limited by toxicity or intolerance) - Subjects' doses of nonsteroidal antiinflammatory drugs (NSAIDs) and oral corticosteroids (less than or equal to 10 mg/day of prednisone or equivalent) must have been kept stable for 4 weeks prior to enrollment.

Doses of 10 mg/day prednisone or equivalent should not be exceeded during the study Exclusion Criteria: - ACR functional class IV or ARA anatomical stage IV - Subjects that are scheduled for surgery or being evaluated for surgery for hands, wrist and feet - Felty's syndrome - Any poorly controlled, clinically significant systemic disease (e.g., chronic obstructive pulmonary disease, congestive heart failure, stroke, chronic renal failure, liver disease) - Poorly controlled diabetes mellitus (e.g., diabetics with HbA1C greater than 8%, peripheral neuropathy, renal/retinal involvement, or vascular disorders) - Malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix within the past 5 years - Abnormal chest x-ray that is clinically significant or bronchiectasis - Within 12 weeks before date of enrollment any of the following occurrences: presence of serious infection (e.g., requiring hospitalization and/or IV antibiotics), frequent, acute, or chronic infections - History of chronic infection - Recent history (within 24 weeks of enrollment) of drug or alcohol abuse - Known to be positive for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus - Presence of any condition that may compromise the ability of the subject to give informed consent - Planned events (e.g., planned hospitalizations, vacations, etc.) that would interfere with the collection of the required assessments and/or may prevent the subject from completing the study according to protocol - White cell count less than or equal to 3.5 x 10^9/L, a neutrophil count of less than or equal to 2.5 x 10^9/L, or platelet count of less than or equal to 125 x 10^9/L at screening - Hemoglobin less than or equal to 8.0 g/dL at screening - Elevated AST or ALT greater than or equal to 1.5 x the upper limit of normal at screening - Elevated serum creatinine greater than or equal to 1.5 x the upper limit of normal at screening - Received intra-articular or systemic corticosteroid injections within 4 weeks before enrollment - Subjects who have received previous treatment with anti-IL-1ra or anti-TNF therapies (e.g., anakinra, etanercept or infliximab) within 4 weeks prior to enrollment - Subjects who are pregnant or breast-feeding, or plan to become pregnant during the course of the study - Subject (man or woman) is of child bearing potential and not using adequate contraceptive precautions - Known allergy to E. coli derived products - Receiving or has received any investigational drug within the previous 30 days or within 5 half-lives of any investigational drug, whichever is greater (or is currently using an investigational device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
% of subjects continuing Kineret® therapy at the end of the study (I.e., responders according to pre-defined response assessment criteria.)

SECONDARY OUTCOMES:
Change in Health Related Quality of Life (HRQOL) scores at the end of study weeks 12, 24, 36 and 48.
feasibility of simpleject device
treatment response (ACR scores, DAS 28) at the end of study weeks 12, 24, 36 and 48.
Safety of Kineret® when added to current DMARD therapy.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com